CLINICAL TRIAL: NCT07289412
Title: Evaluation of Survival and Clinical Outcomes of Patients Treated With Isolated All-inside Meniscal Sutures or With Meniscal Sutures Associated With Ligament Reconstruction
Acronym: Men Repair
Status: Not yet recruiting | Type: Observational
Sponsor: Stefano Zaffagnini (Other)
Responsible Party: Sponsor-Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: Men Repair
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Suture, Complication; Ligament Laceration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Meniscal tears are among the most common injuries of the knee joint. The average annual incidence is between 60 and 70 cases per 100,000 people. Among young athletes, these injuries account for 20-30% of all knee injuries, while in individuals over 50 they are frequently present even without symptoms (up to 60%). Meniscal tears often coexist with other intra-articular injuries: about one third of all cases occur together with an ACL rupture, which significantly increases the likelihood of a meniscal lesion. Possible treatments range from total meniscectomy, partial or selective meniscectomy, to meniscal suturing.

Compared with meniscectomy, meniscal repair preserves meniscal function and reduces the risk of progression to knee osteoarthritis from 51.42% (after meniscectomy) to 21.28% in patients who undergo meniscal repair. The main meniscal suture techniques are classified as inside-out, outside-in, and all-inside.

The present study aims to analyze the failure rates in patients who underwent meniscal repair using the all-inside technique at a single referral center, evaluating the complication rate, the need for reoperation, and the clinical satisfaction of the operated patients.

The results obtained aim to improve the understanding of the effectiveness of all-inside meniscal sutures-electively used at our referral center-compared with inside-out techniques.

The purpose of this study is to collect and analyze the cases of patients surgically treated with all-inside sutures for isolated meniscal tears or tears associated with other ligament injuries. The goal is to evaluate the survival and reoperation rates in patients who underwent all-inside meniscal repair for isolated meniscal injuries or those associated with ligament injuries, aged between 12 and 65 years, operated on at the II Clinic of the Rizzoli Orthopaedic Institute between 01/01/2017 and 30/06/2025, with a minimum follow-up of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients.
* Patients who underwent meniscal repair surgery using the all-inside technique for isolated meniscal lesions or lesions associated with ligament injuries between 01/01/2017 and 30/06/2025, with a minimum follow-up of two years.
* Patients aged between 12 and 65 years at the time of surgery.
* Patients who have provided consent to participate in the study.
* Patients who underwent preoperative radiological investigations (MRI) of the affected knee showing meniscal lesions requiring surgical treatment, also confirmed during diagnostic arthroscopy.

Exclusion Criteria:

* Meniscal lesions resulting from previous meniscal repairs.
* Patients younger than 12 years or older than 65 years at the time of surgery.
* Patients who did not provide informed consent.
* Patients who are no longer contactable.
* Patients who did not engage in sports activity in the 2 years prior to surgery

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited among both male and female subjects, aged 12 years or older and under 65 years at the time of surgery, who underwent meniscal repair using the all-inside technique for isolated meniscal lesions or lesions associated with other ligament injuries at the II Clinic of the Rizzoli Orthopedic Institute between 01/01/2017 and 30/06/2025. Only patients with a minimum follow-up of 2 years from the date of surgery will be enrolled
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 24 months after surgery
  Failures and reoperations will be recorded and documented within the CRF, during telephone questionnaires, and through the patient's clinical documentation

SECONDARY OUTCOMES:
SPORTS (Subjective Patient Outcome for Return To Sports) Score | 24 months after surgery
  This is a subjective questionnaire that assesses the level of return to sports activity compared to the pre-injury condition through a numerical scale consisting of 0, 3, 6, 9, and 10, accompanied by a verbal evaluation of athletic performance ranging from "disabled," corresponding to "0," to "good," corresponding to "10." These numerical values are arranged in increasing order in accordance with the assessment of return to sports activity relative to pre-injury performance
IMPACT activity level score | 24 months after surgery
  It is an objective rating scale that allows the assessment of the level of impact on the knee based on the type of sport practiced. The different sports activities, according to their impact level, are classified as "Low," "Intermediate," and "High." This makes it possible to evaluate the impact level before and after surgery by comparing the type of sports activity performed by the patient prior to and following the surgical procedure
Lysholm Knee Score | 24 months after surgery
  It is a validated measurement scale that assesses knee function through 8 items that allow the evaluation of the knee's condition in response to the functional demands of daily living activities. This assessment tool is used to evaluate surgical outcomes in patients undergoing procedures for ligament or meniscal knee injuries. The final score is obtained by summing the points from the various items and ranges from 0 to 100. The scores are divided into subgroups: Excellent (95-100); Good (84-94); Fair (65-83); Poor (<64)
Tegner Score | 24 months after surgery
  It allows the estimation of a subject's level of physical activity with a score ranging from 0 to 10, where 0 represents 'disability' and 10 represents 'participation in competitive sports, such as football at the national or international level.' This score is the most commonly used to define the activity level of patients with knee disorders. In the study, the Tegner Score will be completed directly by the investigator through an interview with the patient
VAS (Visual Analog Scale) | 24 months after surgery
  It is a unidimensional quantitative 10-point numerical scale for pain assessment, represented by a 10 cm horizontal line without visible numerical markings, with the two ends labeled "no pain" (0) and "worst possible pain" (10). The patient is asked to mark a point on the line that represents the intensity of pain perceived at that moment. The investigator then measures the distance from the "0" point to quantify the pain. This scale will also be used to assess pre- and postoperative pain at the lateral compartment of the knee. This data will help evaluate the onset of pain following surgery at the site of placement of the metal chambers used for graft fixation in lateral tenodesis. Pain in the lateral femorotibial compartment reported as greater than 2 on the VAS scale will be considered as the presence of pain in the lateral compartment, while a value less than or equal to 2 will be considered as the absence of pain in the lateral compartment of the knee
KOOS (Knee Injury and Ostearthritis Outcome Score) score | 24 months after surgery
  It is a subjective score composed of 42 questions divided into 5 main domains. These domains investigate different aspects of symptoms, daily activities, and knee-related quality of life, and are divided as follows:
  * Symptoms: 7 questions, 2 regarding stiffness;
  * Pain: 9 questions;
  * Function and activities of daily living: 17 questions;
  * Sport and recreational activities: 5 questions;
  * Knee-related quality of life: 4 questions; All questions use the same response format, employing a quantitative scale from 0 (no problem) to 4 (severe difficulty). Scores are calculated separately for each domain and converted into a percentage score, where 100 represents excellent physical condition with no symptoms, and 0 represents severe disability with limitations in daily activities and constant symptoms even at rest.
International Knee Documentation Committee (IKDC) | 24 months after surgery
  The IKDC form is a subjective knee evaluation tool that assesses the limitations a subject may experience in daily and sports activities, as well as the presence or absence of symptoms. The IKDC assessment consists of three main domains: Symptoms: including pain, stiffness, swelling, and feelings of locking; Sport and daily activities; Current knee function and function prior to injury.
  The questionnaire comprises 10 questions: seven items assess the patient's symptoms, one item addresses sports participation, one item-composed of 9 points-evaluates the difficulties the patient experiences in performing daily living activities, and the final item measures the current knee function.
  The score ranges from 0 to 100, with 100 representing no limitations or symptoms, indicating an excellent outcome. The further the score deviates from 100, the worse the result. Scores can be categorized into four groups: excellent (80-100), good (60-80), fair (30-60), and poor (0-30)
Number of Participants with Radiological Assessment | 24 months after surgery
  Imaging materials available to the patient will be collected. And which one performed at a minimum follow-up of two years, already completed and in the patient's possession at the time of study participation, will be analyzed. The level of meniscal tissue healing will be assessed, and cartilage damage will be quantified using the ICRS Cartilage Score

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy